CLINICAL TRIAL: NCT05353725
Title: Extracorporeal Membrane Oxygenation in COVID-19, Influenza and ARDS of Other Ethiologies
Brief Title: Extracorporeal Membrane Oxygenation in Coronavirus Disease (COVID-19), Influenza and ARDS of Other Ethiologies
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jernej Berden, MD, PhD, Deputy Head of Department of Internal Intensive Care Medicine, University Medical Centre Ljubljana
Other Study IDs: ECMO in ARDS
Record Dates: First submitted 2022-04-28; First posted 2022-04-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: ARDS; COVID-19; Influenza
Keywords: Extracorporeal Membrane Oxygenation; ARDS; COVID-19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 ARDS: Patients with COVID-19 ARDS on veno-venous ECMO (vvECMO)
- Influenza ARDS: Patients with Influenza ARDS on vvECMO
- ARDS of Other Ethiologies: Patients with ARDS of Other Ethiologies on vvECMO

SUMMARY:
A comparison of clinical characteristics and outcomes of patients on extracorporeal membrane oxygenation (ECMO) in COVID-19, influenza and ARDS of other ethiologies

DETAILED DESCRIPTION:
All ARDS patients on extracorporeal membrane oxygenation (ECMO) during January 1st 2016 and January 10th 2022 in University Medical Center Ljubljana were included and their clinical characteristics and outcomes were studied according to ARDS ethiology: COVID-19, influenza and other ethiologies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute respiratory distress syndrome (ARDS) on extracorporeal membrane oxygenation (ECMO)
* 18 years or older

Exclusion Criteria:

* Patient not eligible for ECMO treatment per institutional guidelines (terminal illness, palliative care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory distress syndrome (ARDS) on extracorporeal membrane oxygenation (ECMO)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
180-day survival | From day of ECMO-implant for every 24 hours until date of death or survival at 180 days
  180-day survival from ECMO implantation

SECONDARY OUTCOMES:
Days on ECMO | From day of ECMO-implant for every 24 hours until date of weaning or death
  Days on ECMO from ECMO implantation
Weaning from ECMO | From day of ECMO-implant until date of death or weaning
  Weaning from ECMO
ICU length of stay | From day of ICU-admission for every 24 hours until date of death or date of ICU discharge
  ICU length of stay from ECMO implantation
ICU survival | From day of ICU-admission for every 24 hours until date of death or survival at ICU discharge
  ICU survival from ECMO implantation
Hospital survival | From day of hospital admission for every 24 hours until date of death or survival at hospital discharge
  Hospital survival from ECMO implantation
30-day survival | From day of ECMO-implant for every 24 hours until date of death or survival at 30 days
  30-day survival from ECMO implantation
90-day survival | From day of ECMO-implant for every 24 hours until date of death or survival at 90 days
  90-day survival from ECMO implantation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanelli V, Giani M, Grasselli G, Mojoli F, Martucci G, Grazioli L, Alessandri F, Mongodi S, Sales G, Montrucchio G, Pizzi C, Richiardi L, Lorini L, Arcadipane A, Pesenti A, Foti G, Patroniti N, Brazzi L, Ranieri V. Extracorporeal membrane oxygenation for COVID-19 and influenza H1N1 associated acute respiratory distress syndrome: a multicenter retrospective cohort study. Crit Care. 2022 Feb 5;26(1):34. doi: 10.1186/s13054-022-03906-4. PMID 35123562
- [Background] Chong WH, Saha BK, Medarov BI. A systematic review and meta-analysis comparing the clinical characteristics and outcomes of COVID-19 and influenza patients on ECMO. Respir Investig. 2021 Nov;59(6):748-756. doi: 10.1016/j.resinv.2021.07.006. Epub 2021 Aug 17. PMID 34481816
- [Background] Blazoski CM, Baram M, Yang Q, Hirose H. Outcomes of extracorporeal membrane oxygenation in influenza versus COVID-19 during the first wave of COVID-19. J Card Surg. 2021 Oct;36(10):3740-3746. doi: 10.1111/jocs.15888. Epub 2021 Aug 9. PMID 34369601